CLINICAL TRIAL: NCT01337154
Title: A Randomized, Placebo-Controlled Phase 2b Study of Tamibarotene Plus Paclitaxel and Carboplatin Versus Placebo Plus Paclitaxel and Carboplatin as First Line Treatment for Subjects With Advanced Non-Small Cell Lung Cancer
Brief Title: First Line Study of Tamibarotene in Combination for Advanced Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Interim analysis showed that the primary endpoint would not be met.
Sponsor: CytRx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAMI-P2-NSCLC-01
Record Dates: First submitted 2011-04-15; First posted 2011-04-18 (Estimated); Last update posted 2013-06-28 (Estimated); Status verified 2013-06

CONDITIONS: Stage IIIB Non-small Cell Lung Cancer With Pleural Effusion; Stage IV Non-small Cell Lung Cancer
Keywords: NSCLC; non-small cell lung cancer; tamibarotene
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — tamibarotene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tamibarotene (Experimental): Subjects will receive tamibarotene, 6 mg/m2, divided as twice daily orally starting 1 week before chemotherapy and continuing through all 6 cycles and through the duration of the study. Chemotherapy will include paclitaxel (IV; 200 mg/m2) and carboplatin (IV; AUC=6)administered once every 3 weeks for up to 6 cycles.
  Interventions: Drug: Tamibarotene
- Placebo (Placebo Comparator): Subjects will take an equal number of placebo tablets as the group receiving tamibarotene divided as twice daily orally, starting 1 week before chemotherapy and continuing through all 6 cycles and through the duration of the study. Paclitaxel (IV; 200 mg/m2) and carboplatin (IV; AUC=6) will be administered once every 3 weeks for up to 6 cycles.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tamibarotene — Tablet, 6 mg/m2, oral, divided into twice a day dosing.
  Arms: Tamibarotene
Drug: Placebo — Tablets, orally, daily
  Arms: Placebo

SUMMARY:
The goal of this study is to determine the progression-free survival and objective response rate in subjects with either stage IIIB with pleural effusion NSCLC or stage IV NSCLC who are treated with up to six cycles of paclitaxel plus carboplatin and either tamibarotene or placebo. Subjects will be randomly assigned to receive tamibarotene, 6 mg/m2, divided as twice daily orally, or an equal number of matching placebo tablets, starting 1 week before chemotherapy and continuing through all 6 cycles and beyond. Subjects will be assessed for response on Day 50, Day 113, then every other month using the Response Evaluation Criteria in Solid Tumors (RECIST 1.1).

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be at least 18 years of age
* Subjects must have pathological findings consistent with primary non-small cell lung cancer of any histology.
* Subjects must have either stage IIIB with pleural effusion or IV NSCLC with radiographically measurable disease (RECIST 1.1 criteria). Women non-smokers with stage IV NSCLC should be screened for EGFR mutation and if positive be excluded from the study and placed on an EGFR kinase inhibitor.
* Subjects must have an ECOG Performance Status ≤2.
* If corticosteroids are required for controlling cerebral edema, subjects must be on a stable dose for at least 1 week.
* Subjects must have recovered from any toxicity of prior therapies.
* Subjects must be at least 4 weeks removed from surgery or radiation therapy.
* Subjects must have a life expectancy of at least 12 weeks.
* Subjects must have adequate bone marrow function (defined as an absolute neutrophil count of ≥1500 cells/mm3 and platelet count ≥100,000 cells/mm3), liver function with total bilirubin ≤2.0 mg/dL, and serum creatinine ≤1.5 x institutional ULN.
* Subjects must be able to understand and be willing to sign a written informed consent document.
* Tamibarotene, as with all retinoids, is teratogenic. Therefore, female subjects of childbearing potential must agree to use 2 effective methods of contraception (hormonal, barrier method of birth control, or abstinence) and sexually-active male subjects must agree to use an effective method of contraception (hormonal or barrier method of birth control or abstinence) while participating in this study and for six months afterwards. Women of childbearing potential must have a negative pregnancy test ≤1 week prior to registration.
* Subjects must be able to swallow tablets.
* If available, tumor specimens must be submitted for immunohistochemistry analyses with their pathology reports.

Exclusion Criteria:

* Subjects who have received or are currently receiving chemotherapy or antibody therapy, or are enrolled in another treatment clinical trial.
* Subjects with a coagulopathy or bleeding disorder.
* Clinically evident congestive heart failure >class II of the New York Heart Association (NYHA) guidelines.
* Serious, clinically significant cardiac arrhythmias, defined as the existence of an absolute arrhythmia or ventricular arrhythmias classified as Lown III, IV or V.
* History or signs of active coronary artery disease with or without angina pectoris (i.e. myocardial infarction with 6 months prior to enrollment, uncontrolled angina, electrocardiographic evidence of acute ischemia).
* Subjects who have a serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol or may not be able to comply with the safety monitoring requirements of the study.
* HIV-positive subjects; however, subjects will not be routinely screened for HIV.
* Subjects who are allergic to any of the intended chemotherapies.
* Female subjects who are pregnant or breast-feeding.
* Active, clinically significant serious infection requiring treatment with antibiotics, antivirals, or antifungals.
* Subjects with peripheral neuropathy ≥grade 2
* Prior systemic treatment for locally advanced or metastatic disease (exception below): Prior adjuvant chemotherapy for Stage I-III or combined modality chemotherapy-radiation for locally advanced disease allowed if completed >12 months prior to randomization.
* Subjects with brain metastases are only eligible if treated and neurologically stable with no ongoing requirement for corticosteroids, e.g., dexamethasone, for at least 2 weeks.
* Subjects with hypertriglyceridemia (>1000 mg/dL).
* Subjects with elevated liver function tests if AST is ≥2.5x the institutional or central laboratory's upper limit of normal for subjects without liver metastases, or >5x the institutional or central laboratory's upper limit of normal for subjects with liver metastases.
* Subjects with HbA1c ≥8.0.
* Subjects taking vitamin A either as a supplement or as part of a multivitamin unless there has been at least a 2 week washout.
* Subjects using concomitant medications that are known inducers or inhibitors of CYP3A4 up to 14 days before Cycle 1 Day 1 (pimozide, diltiazem, erythromycin, clarithromycin, and quinidine, and amiodarone) should be excluded from the study.
* Subjects whose tumors cannot be adequately measured per RECIST 1.1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2011-04; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | Within 18 months of study start.
  Progression-free survival (PFS) is defined as the time from enrollment (i.e., assignment of subject ID number) to first documentation of objective tumor progression or to death due to any cause in the absence of previous documentation of objective tumor progression.

SECONDARY OUTCOMES:
Objective response rate | Within 18 months of study start.
  Objective tumor response will be evaluated using the RECIST 1.1 criteria.
Overall survival | Within 24 months of study start.
Assessment of quality of life | Within 24 months of study start.
  EORTC QLQ-C30 version 3.

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Arrieta, M.D., Principal Investigator — Instituto Nacional de Cancerologia, Columbia
Locations (26):
- United States (3):
  - Desert Hematology Oncology Medical Group, Inc., Rancho Mirage, California
  - Kansas City Cancer Center, Kansas City, Kansas
  - Hackensack University Medical Center, Hackensack, New Jersey
- Bulgaria (3):
  - Department of Medical Oncology, Specialized Hospital for Active Treatment of Oncological Diseases, Sofia
  - Medical Oncology Clinic, Multiprofile Hospital for Active Treatment, Varna
  - Department of Medical Oncology, Complex Oncology Center, Veliko Tarnovo
- India (8):
  - NIZAM's Institute of Medical Sciences, Hyderabad, Andhra Pradesh
  - M S Patel Cancer Centre, Shree Krishna Hospital, Anand, Gujarat
  - Curie Manavata Cancer Centre, Nashik, Maharashtra
  - Shatabdi Super Speciality Hospital, Nashik, Maharashtra
  - Noble Hospital, Pune, Maharashtra
  - Dr. Kamakshi Memorial Hospital, Chennai, Pallikaranai
  - G Kuppuswamy Naidu Memorial Hospital, Valvadi Narayanaswamy Cancer Centre, Coimbatore, Pappanaickenpalayam
  - Orchid Nursing Home, Kolkata, West Bengal
- Instituto Nacional de Cancerologia, Mexico City, Mexico
- Russia (5):
  - State Medical Institution: Arkhangelsk Regional Clinical Oncology Center, Arkhangelsk
  - State Therapeutical and Prophylatic Institution: Chelyabinsk Regional Clinical Oncology Center, Chelyabinsk
  - State Medical Instituion Kursk Regional Oncology Center, Kursk
  - Non-State Medical Institution: Central Clinical Hospital #2, Moscow
  - St. Petersburg State Healthcare Institution: City Clinical Oncology Center, Saint-Pertersburg
- Ukraine (6):
  - Public Institution: Dnipropetrovsk City Multispeciality Clinical Hospital #4, Dnipropetrovsk
  - Public Clinical Treatment and Prophylaxis Instituion: Donetsk Regional Antitumor Center, Donetsk
  - Ivano-Frankivsk Regional Oncology Center, Ivano-Frankivsk
  - Public Healthcare Instituion: Kharkiv Regional Clinical Oncology Center, Kharkiv
  - Kyiv City Clinical Oncology Center, Kyiv
  - Zakarpattia Regional Clinical Oncology Center, Uzhhorod